CLINICAL TRIAL: NCT03990623
Title: To Evaluate Perfusion Changes to the Liver Following Pre-Operative Portal Vein Embolization for Patients With Liver Cancer
Brief Title: CT Perfusion Scans in Detecting Changes in Blood Flow to the Liver After Portal Vein Embolization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-0399; NCI-2019-02648 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0399 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2019-06-17; First posted 2019-06-19 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2022-09

CONDITIONS: Liver and Intrahepatic Bile Duct Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Cytidine Triphosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (CT perfusion scans, liver biopsy) (Experimental): Prior to PVE, patients undergo CT perfusion scan of the liver and liver biopsy over 15 minutes. Patients undergo a second CT perfusion scan immediately after PVE and a third CT perfusion scan 3-6 weeks post PVE.
  Interventions: Radiation: Computed Tomography Perfusion Imaging; Procedure: Liver Biopsy

INTERVENTIONS:
Radiation: Computed Tomography Perfusion Imaging — Undergo perfusion CT
Procedure: Liver Biopsy — Undergo liver biopsy
  Other Names: Biopsy of Liver

SUMMARY:
This trial studies the use of computed tomography (CT) perfusion scans in detecting changes in blood flow to the liver after portal vein embolization in patients with liver cancer. CT perfusion scans use a standard contrast drug given by vein to measure blood flow to the liver. CT perfusion scans may predict the rate and amount of growth of new, healthy tissue on one side of the liver after a portal vein embolization and detect change to the size of the liver tumor as result of the procedure.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess whether perfusion changes to the liver following portal vein embolization (PVE) correlate with hypertrophy of the future liver remnant (FLR).

SECONDARY OBJECTIVES:

I. To assess perfusion changes to liver tumors following PVE. II. To assess whether PVE may affect tumor growth.

OUTLINE:

Prior to PVE, patients undergo CT perfusion scan of the liver and liver biopsy over 15 minutes. Patients undergo a second CT perfusion scan immediately after PVE and a third CT perfusion scan 3-6 weeks post PVE.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned to undergo major liver resection for cancer who need PVE to increase the size of the FLR prior to surgery.
* Patients who are able to understand and give consent to participate in the study.

Exclusion Criteria:

* Pregnant or nursing.
* Allergy to iodinated contrast which cannot be safely pre-medicated.
* History of severe renal dysfunction (glomerular filtration rate [GFR] < 30 mL/min/1.73 square meters). Patients with a GFR between 30-50 mL/min/1.73 square meters will receive the standard contrast-induced nephropathy prophylaxis at our institution (i.e. N-acetylcysteine and sodium bicarbonate [150 mEq/L] in D5W intravenous).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2018-07-21 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Perfusion changes to the liver following portal vein embolization (PVE) | Baseline up to 6 weeks post PVE
  Will assess whether perfusion changes to the liver following PVE correlate with hypertrophy of the future liver remnant (FLR). Perfusion and FLR hypertrophy are two continuous variables. Each patient will serve as his/her own control. Perfusion to the liver (1) before PVE, (2) immediately after PVE, and (3) 3-6 weeks following PVE will be measured and compared. The changes in perfusion will be compared with FLR hypertrophy at the 3-6 week time point to assess correlation.

SECONDARY OUTCOMES:
Changes to tumor cellular proliferation following PVE | Baseline up to 6 weeks post PVE
  Will assess perfusion changes to liver tumors following PVE and whether this may affect tumor growth kinetics. Each patient will serve as his/her own control. Perfusion to the liver tumor(s) (1) before PVE, (2) immediately after PVE, and (3) 3-6 weeks following PVE will be measured and compared. Since a percutaneous biopsy will be performed of a single liver tumor before PVE and the tumor explant will be available following surgical resection, changes to tumor cellular proliferation following PVE can be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Y Huang, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org